CLINICAL TRIAL: NCT03032523
Title: Detecting Neonatal Hypoglycemia Using Real-Time Continuous Glucose Monitoring (CGM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura Nally, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 36668
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Monitoring CGM Group (Experimental): Participants wear a CGM that is blinded at bedside (to participant and clinical staff) but remotely monitored by study staff. If a blood sugar less than 46 mg/dl occurs, the study staff receive a notification and ask the clinical staff to perform a confirmation standard of care glucose test.
  Interventions: Diagnostic Test: Standard of care glucose test
- Blinded CGM Group (No Intervention): Participants wear a blinded CGM during the study period. Values are blinded to study staff, participant, and clinical staff.

INTERVENTIONS:
Diagnostic Test: Standard of care glucose test — If the CGM in the remote monitoring group detects a blood sugar less than 46mg/dl, a confirmatory standard of care glucose test will be performed to confirm the low blood sugar.
  Arms: Remote Monitoring CGM Group

SUMMARY:
Hypoglycemia is the most common metabolic problem faced after birth. The investigators will be studying the utility of using a continuous glucose monitoring(CGM) system to more closely monitor low blood sugars in newborns. The investigators will evaluate the number of hypoglycemic events detected using CGM and compare it to those detected using current standard of care screening methods.

DETAILED DESCRIPTION:
A CGM will be subcutaneously inserted by trained staff on a healthy area of skin and will be calibrated according to the manufacturer's instructions. Blood glucose measurements will be taken using a blinded study glucometer to calibrate the device. Calibration by trained study staff will take place about every 12 hours. Sensor insertion sites will be monitored for infection throughout the course of the study by nursing and clinical staff or by trained study staff on an as needed basis. At the conclusion of the study, the CGM will be removed and assessed for signs of infection. Study duration will be up to 7 days while the patient is admitted to the hospital.

Participants will be randomized into 2 groups. The control group will have a blinded CGM in place for the duration of the study. The remote monitoring group will be blinded to clinical staff. This group will have a CGM connected to an iPod that sends continuous glucose data to the study phone and will be monitored 24/7 by study staff. If a blood sugar level of <46 mg/dl is detected, the infant will first be evaluated for positioning that could be causing a falsely low value. If the infant is re-positioned and CGM continues to show a blood sugar level of <46 mg/dl, study staff will prompt the nurse taking care of the patient to obtain a capillary glucose value to verify the low blood sugar and treat it as deemed appropriate by the clinical team.

The investigators will evaluate the number of hypoglycemic events that occur in the blinded CGM group versus the number that occur in the remote monitoring group to assess if the CGM is able to more sensitively detect low blood sugars in infants than current hospital standard of care measures.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are at least 34 weeks gestation that are born to mothers with gestational or pre-gestational diabetes and are admitted to LPCH are eligible for the study.

Exclusion Criteria:

* Infants <2,000 grams will be excluded from the study. Infants will also be excluded if they have an anomaly of the skin or subcutaneous tissue that would prevent proper adhesion, placement, and function of the sensor.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Nally, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers attending obstetrics clinics at Stanford University were approached if they met inclusion criteria. 119 mothers were approached, 66 declined to participate, 23 were lost to follow up after initially discussing the study, 6 were unable to participate because research staff were not available at the time of birth, and 3 were ineligible.
Groups:
- Remote Monitoring CGM Group: Participants wear a CGM that is blinded at bedside (to participant and clinical staff) but remotely monitored by study staff. If a blood sugar less than 46 mg/dl occurs, the study staff receive a notification and ask the clinical staff to perform a confirmation standard of care glucose test.
  Standard of care glucose test: If the CGM in the remote monitoring group detects a blood sugar less than 45 mg/dl, a confirmatory standard of care glucose test will be performed to confirm the low blood sugar.
Period: Overall Study
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group
Started | 15 | 6
Completed | 12 | 4
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All infants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Customized [Count of Participants; unit: Participants]
  Less than 24 hours of life | 14 | 6 | 20
  24-48 hours of life | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 2 | 10
  Asian | 3 | 2 | 5
  Pacific Islander | 0 | 1 | 1
  Other | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Sensor-detected Hypoglycemia
Description: Reported values in the table represent the cumulative number of hypoglycemic events detected by the sensor that were not detected by the hospital standard of care measures across all participants.
Time Frame: up to 8 days
Population: Participants in the remote monitoring group were eligible for analysis. 3 were excluded from the remote monitoring group for the analysis. Blinded CGM participants did not have a verification glucose check, thus sensor-detected hypoglycemia was not verified, and thus were not reported in the analysis.
Measure: Number; unit: events
Groups:
- Remote Monitoring CGM Group: Participants wear a CGM that is blinded at bedside (to participant and clinical staff) but remotely monitored by study staff. If a blood sugar less than 46 mg/dl occurs, the study staff receive a notification and ask the clinical staff to perform a confirmation standard of care glucose test.
  Standard of care glucose test: If the CGM in the remote monitoring group detects a blood sugar less than 45mg/dl, a confirmatory standard of care glucose test will be performed to confirm the low blood sugar.
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group
Number analyzed (Participants) | 12 | 0
events
  Hypo Events Detected by Sensor (not SOC) | 5 |
  Hypo Events Detected by SOC and not sensor | 1 |

2. Secondary Outcome: Sensitivity of the CGM to Detect Hypoglycemia.
Description: True positive rate.
Time Frame: up to 7 days
Population: Participants in the Remote Monitoring CGM Group were analyzed. 3 were excluded from the remote monitoring group for the analysis. Those in the blinded group were unable to be analyzed because the CGM was blinded and did not prompt a BG check.
Measure: Number; unit: % of true hypoglycemic events
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group
Number analyzed (Participants) | 12 | 0
% of true hypoglycemic events | 86 |

3. Secondary Outcome: Specificity of CGM to Detect Hypoglycemic Events
Description: True negative rate
Time Frame: up to 7 days
Population: 12 participants had sensor data for analysis. 3 were excluded from the remote monitoring group for the analysis. Blinded CGM participants did not have a verification glucose check, thus specificity could not be calculated on these participants.
Measure: Number; unit: % of true negative events
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group
Number analyzed (Participants) | 12 | 0
% of true negative events | 91 |

ADVERSE EVENTS:
Time Frame: Up to 7 days of life
Description: Sensor sites on infants examined twice daily by research staff and daily chart reviews were performed.
Groups:
- Remote Monitoring CGM Group: Participants wear a CGM that is blinded at bedside (to participant and clinical staff) but remotely monitored by study staff. If a blood sugar less than 45 mg/dl occurs, the study staff receive a notification and ask the clinical staff to perform a confirmation standard of care glucose test.
  Standard of care glucose test: If the CGM in the remote monitoring group detects a blood sugar less than 46mg/dl, a confirmatory standard of care glucose test will be performed to confirm the low blood sugar.
Arm/Group | Remote Monitoring CGM Group | Blinded CGM Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 1/15 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Monitoring CGM Group (N=15) | Blinded CGM Group (N=6)
Retained sensor wire (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One infant retained the sensor wire upon removal of the sensor, which is a very rare, but known risk. No medical intervention related to the retained sensor wire was required.

LIMITATIONS AND CAVEATS:
Because we were unable to recruit 40 infants during the time frame of the randomized trial, we modified the study design to test the additional benefit of using CGM monitoring to detect hypoglycemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03032523/Prot_SAP_000.pdf